CLINICAL TRIAL: NCT04929509
Title: Effectiveness of Self-assembling Peptide (P11-4) and Nano-silver Fluoride Varnish in Management of Enamel White Spot Lesions in Young People (Randomized Controlled Clinical Trial)
Brief Title: P11-4 and Nanosilver Fluoride Varnish in Treatment of White Spot Carious Lesions
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hams Hamed Abdelrahman (Other)
Responsible Party: Sponsor-Investigator, Hams Hamed Abdelrahman, Assistant lecturer, Alexandria University
Organization: Alexandria University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: P11-4 in white spot lesions
Record Dates: First submitted 2021-06-15; First posted 2021-06-18 (Actual); Last update posted 2021-06-18 (Actual); Status verified 2021-06

CONDITIONS: White Spot Lesion
MeSH Terms: interventions — Bifluorid 12; Duraflor

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- self-assembling peptide (P11-4) (Experimental): Curodont Repair; Credentis will be applied to the
  white spot lesion at baseline.
  Interventions: Other: self-assembling peptide
- nanosilver fluoride varnish (Active Comparator): (Study group) Nano-silver fluoride varnish will be applied to the
  white spot lesion at baseline.
  Interventions: Other: nanosilver fluoride varnish
- sodium fluoride varnish (Placebo Comparator): (Control group) Fluoride varnish (Duraflor) will be applied to the
  white spot lesion at baseline and 6 months follow up.
  Interventions: Other: sodium fluoride varnish

INTERVENTIONS:
Other: self-assembling peptide — each Curodont Repair applicator unit contains both Curolox technology for guided enamel regeneration and water for activation of the device, each box contains 10 applicators
  Other Names: Curodont repair
  Arms: self-assembling peptide (P11-4)
Other: nanosilver fluoride varnish — The synthesis of aqueous solution of silver nanoparticles will be carried out via the chemical reduction of silver nitrate (1 mL, 0.11 M) with sodium borohydride (0.3 mL, 0.8 M) and chitosan biopolymer (28.7 mL, 2.5 mg/mL) as a stabilizing agent. Sodium fluoride (10,147 ppm of fluorine) will be incorporated at the end of the experiment.
  Arms: nanosilver fluoride varnish
Other: sodium fluoride varnish — 5% sodium fluoride varnish; One ml of fluoride varnish contains 50 mg of sodium fluoride in an alcohol-based suspension of resins.
  Other Names: duraflor
  Arms: sodium fluoride varnish

SUMMARY:
Background: Great efforts have been undertaken for dental caries prevention. Among the recent remineralizing materials, Nano silver fluoride varnish products which are based on nanotechnology have been proposed for "repairing" enamel . Regenerative medicine-based approaches for caries treatment focus on biomimetic remineralization of initial carious lesions as a minimal invasive therapy using Self-Assembling Peptide P11-4 (Curodont Repair) which enhances remineralization of white spot lesions. Purpose of the Study: The aim of this study is to compare clinically and microbiologically the therapeutic effect of Self Assembling Peptide P11-4 (Curodont Repair), nano silver fluoride varnish and 5% fluoride varnish (Duraflor) on remineralization of enamel White Spot Lesions in permanent teeth of adults.

DETAILED DESCRIPTION:
The study will be a randomized controlled double-blinded study conducted on participants aged 10 to 24 years satisfying the inclusion criteria with visible active white spot lesions on buccal surfaces of permanent teeth. Sixty six patients will be randomly allocated into 3 groups of the three materials: study group 1: one application of Curodont Repair, study group 2: one application of Nano-silver fluoride varnish and Control group twice application of Fluoride Varnish (Duraflor).

ELIGIBILITY:
Inclusion Criteria:

1- An age range of 10-24 years ( age of young adolescents and youth as described by the WHO was selected (WHO, 2019). 2. The presence of at least one visible WSL in the buccal surface of permanent teeth with ICDAS II score of 1, or 2. 3. Completion of an informed consent to participate in the study

Exclusion Criteria:

* 1. Patients receiving the following medications: tetracyclines, any other medication known to stain teeth or any medication causing dry mouth and/or limiting salivary flow. 2. Patients receiving any antibiotic within 1 month prior to each saliva sample collection 3. Selected tooth with microcavities or dentinal involvement due to loss of enamel tissues. 4. Selected tooth with a restoration adjacent to the lesions to avoid false- positive readings. 5. Selected tooth with fluoride application < 3 months prior to study treatment. 6. Selected tooth with discolouration, enamel hypoplasia or fluorosis. 7. Patients with multiple cavitations to avoid variability in microbiological analysis.

Ages: 10 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 66 (Estimated)
Dates: Start 2020-12-05 (Actual); Primary Completion 2021-10-05 (Estimated); Study Completion 2022-01-01 (Estimated)

PRIMARY OUTCOMES:
Change in the activity status of lesions scored using ICDAS-LAA | 12 months
  Change in the activity status of lesions scored using ICDAS-LAA from baseline to final follow up.

SECONDARY OUTCOMES:
Change in mean DIAGNOdent readings. | 12 months
  Change in mean DIAGNOdent readings from baseline to each follow up period
Microbial count of mutans streptococci, lactobacilli. | 6 months
  Microbial count of mutans streptococci, lactobacilli.from baseline to each follow up period

CONTACTS AND LOCATIONS:
Overall Officials: Hala A Amer, PHD, Study Director — Alexandria University; Susan M Saleh, PHD, Principal Investigator — Alexandria University; Yara S Selim, PHD, Principal Investigator — Alexandria University; Sara M Atteya, PHD, Principal Investigator — Alexandria University
Locations (1):
- Faculty of dentistry, Alexandria, Egypt

REFERENCES:
- [Derived] Atteya SM, Amer HA, Saleh SM, Safwat Y. The effect of nano silver fluoride, self-assembling peptide and sodium fluoride varnish on salivary cariogenic bacteria: a randomized controlled clinical trial. Clin Oral Investig. 2024 Feb 23;28(3):167. doi: 10.1007/s00784-024-05562-0. PMID 38388987
- [Derived] Atteya SM, Amer HA, Saleh SM, Safwat Y. Self-assembling peptide and nano-silver fluoride in remineralizing early enamel carious lesions: randomized controlled clinical trial. BMC Oral Health. 2023 Aug 19;23(1):577. doi: 10.1186/s12903-023-03269-4. PMID 37598194